CLINICAL TRIAL: NCT00292877
Title: The Effects of a Humanized Anti-IL-5 Monoclonal Antibody (SB-240563) on Asthma Control, Airway Eosinophilia and the Degree to Which Corticosteroid Treatment Can be Reduced to Maintain Control
Brief Title: The Prednisone-sparing Effect of Anti-IL-5 Antibody (SB-240563)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RP#02-2115; SB-240563/046; 9427-F2453-21C
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: 1. Eosinophilic bronchitis, 2. Asthma, 3. Steroid dependent asthma, 4. Sputum eosinophils, 5. SB-240563 (Mepolizumab)
MeSH Terms: conditions — Asthma | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB-240563 (Mepolizumab)

SUMMARY:
The purpose of this study is to determine if treatment with anti-IL-5 antibody has a prednisone-sparing effect in patients with symptomatic eosinophilic bronchitis (with or without asthma).

DETAILED DESCRIPTION:
Eosinophilic bronchitis, which is identified by quantitative sputum cell counts (eosinophils greater than 2%) is responsive to corticosteroid treatment. It occurs alone or in association with asthma or in some patients with chronic obstructive pulmonary disease (COPD). In most patients the eosinophilic bronchitis responds to treatment with inhaled steroids but in some it requires a minimum dose of prednisone to keep it controlled. At present, there is no outstanding drug which can have a prednisone-sparing effect.

Interleukin (IL)-5 is a cytokine specifically focused on the development, differentiation, recruitment, activation and survival of the eosinophil. The specificity of IL-5 has raised the possibility that blocking it's activity, using humanized monoclonal antibodies, may be useful therapy for eosinophilic bronchitis. Such an antibody (SB-240563) has been introduced for clinical trial. The investigators will compare its effect versus placebo in patients with prednisone-dependant symptomatic eosinophilic bronchitis (with or without asthma) before and after a reduction in prednisone dose to identify if it has a prednisone-sparing effect.

The study is divided into 3 sequential study periods. Period 1: symptomatic eosinophilic bronchitis (with or without asthma) on the same dose of prednisone for 6-weeks or more. Period 2: standardized prednisone reduction (and inhaled steroid if prednisone is discontinued during the study treatment) at intervals of 4-weeks until there is a clinical and eosinophilic exacerbation or bothersome steroid withdrawl effects. Period 3: washout.

The patients will be seen every 2 weeks. Intravenous injections of SB-240563 750mg or placebo will be given at weeks 2,6,10,14 and 18. Doses of prednisone will be reduced in a standard way.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, aged 18-70 years, who have been followed as an outpatient and who have been found to require a minimum dose of prednisone treatment (in addition to high-dose inhaled steroid treatment) to prevent frequent exacerbations associated with induced sputum eosinophilia.
2. Patients will be enrolled if, at screening and baseline visits, they demonstrate sputum eosinophilia and symptoms. The symptoms may effect activity and sleep but should not, in the opinion of the treating physician, be severe enough to be of concern.
3. While FEV1 after withholding bronchodilators appropriately, before and after inhaled salbutamol (200 mg), and methacholine PC20 will be measured, these need not be abnormal since the prednisone is required for the control of eosinophilic bronchitis and any clinical consequences of this, and because the bronchitis can occur without these features of asthma.
4. On the same doses of corticosteroids for a least one-month.

Exclusion Criteria:

1. Pregnancy, breast-feeding or lack of effective contraception in females of childbearing potential or females who are postmenopausal <1 year.
2. Baseline FEV1 before bronchodilator of 40% or less of predicted. This lower FEV1 is acceptable since chronic airflow limitation secondary to the eosinophilic bronchitis or asthma is not an exclusion criteria. Neither is current or ex-cigarette smoking providing that the best FEV1 in these patients has been >60% predicted normal or the best FEV1/VC ratio has been >60% in the past two years.
3. Exposure to a relevant seasonal environmental allergen, known to worsen asthma control, during the study period.
4. Respiratory tract infection in the 4-weeks before the baseline visit.
5. Clinical exacerbation requiring extra prednisone treatment in the 4-weeks before V1.
6. Other cardiac, pulmonary, renal or systemic diseases that in the investigator's opinion may interfere with the study results or compromise subject's safety.
7. Previous participation in any study using anti-monoclonal drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-01; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The prednisone-sparing effect of SB-240563 versus placebo as
indicated by the absolute and percentage dose reduction possible without a clinical exacerbation (as measured by the Juniper ACQ in patients with asthma or by Likert symptom scores +/- FEV1 in patients with eosinophilic bronchitis without asthma).

SECONDARY OUTCOMES:
The prednisone-sparing effect of SB-240563 or placebo as indicated
by the absolute and percentage dose reduction possible without a clinical
exacerbation as measured by
a.% sputum eosinophils, b. FEV1 % predicted and methacholine PC20., c. Blood eosinophils, d. Amount of rescue salbutamol use., e. Time to exacerbation.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick E Hargreave, MD, Principal Investigator — McMaster University
Locations (1):
- Firestone Institute for Respiratory Health, St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Sanderson CJ. The biological role of interleukin 5. Int J Cell Cloning. 1990 Jan;8 Suppl 1:147-53; discussion 153-4. doi: 10.1002/stem.5530080713. PMID 2182734
- [Background] Leckie MJ, ten Brinke A, Khan J, Diamant Z, O'Connor BJ, Walls CM, Mathur AK, Cowley HC, Chung KF, Djukanovic R, Hansel TT, Holgate ST, Sterk PJ, Barnes PJ. Effects of an interleukin-5 blocking monoclonal antibody on eosinophils, airway hyper-responsiveness, and the late asthmatic response. Lancet. 2000 Dec 23-30;356(9248):2144-8. doi: 10.1016/s0140-6736(00)03496-6. PMID 11191542
- [Background] Djukanovic R, Roche WR, Wilson JW, Beasley CR, Twentyman OP, Howarth RH, Holgate ST. Mucosal inflammation in asthma. Am Rev Respir Dis. 1990 Aug;142(2):434-57. doi: 10.1164/ajrccm/142.2.434. PMID 2200318
- [Background] Djukanovic R, Sterk PJ, Fahy JV, Hargreave FE. Standardised methodology of sputum induction and processing. Eur Respir J Suppl. 2002 Sep;37:1s-2s. doi: 10.1183/09031936.02.00000102. No abstract available. PMID 12361359
- [Background] Pavord ID, Brightling CE, Woltmann G, Wardlaw AJ. Non-eosinophilic corticosteroid unresponsive asthma. Lancet. 1999 Jun 26;353(9171):2213-4. doi: 10.1016/S0140-6736(99)01813-9. No abstract available. PMID 10392993
- [Derived] Nair P, Pizzichini MM, Kjarsgaard M, Inman MD, Efthimiadis A, Pizzichini E, Hargreave FE, O'Byrne PM. Mepolizumab for prednisone-dependent asthma with sputum eosinophilia. N Engl J Med. 2009 Mar 5;360(10):985-93. doi: 10.1056/NEJMoa0805435. PMID 19264687